CLINICAL TRIAL: NCT03470389
Title: Establishment and Assessment of the HVPG Using Biofluid Mechanics (HVPGBFM)
Acronym: HVPGBFM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiayun Lin, Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JYLJ021
Record Dates: First submitted 2018-02-25; First posted 2018-03-19 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Liver Cirrhosis; Hypertension, Portal
Keywords: Liver Cirrhosis; Hypertension, Portal; Hepatic Venous Pressure Gradient (HVPG); Biofluid Mechanics; Noninvasive
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HVPG (Experimental): Each patient's computed tomography, blood tests, Doppler ultrasound and HVPG measurement will be performed within 30 days and treatments that may affect HVPG value will be avoided during this period.
  Interventions: Procedure: HVPG measurement

INTERVENTIONS:
Procedure: HVPG measurement — Each patient's computed tomography, blood tests, Doppler ultrasound and HVPG measurement will be performed within 30 days and treatments that may affect HVPG value will be avoided during this period.
  Other Names: Blood test; Doppler ultrasound; Computed tomography

SUMMARY:
This study is a prospective, non-controlled, multicentre trial in patients with cirrhosis or portal hypertension. In this study, the investigators aim to establish the HVPG using biofluid mechanics (HVPGBFM) model using biofluid mechanics methods and validate the HVPGBFM model. A total of 200 patients will be recruited in this study and each patient will undergo computed tomography, blood tests, Doppler ultrasound and HVPG measurement. The study consists of two independent and consecutive cohorts: original cohort (100 patients) and validation cohort (100 patients). The researchers will establish and improve the HVPGBFM model in the original cohort and assess the model in the validation cohort.

DETAILED DESCRIPTION:
Consecutive patients are randomly assigned 1:1 to either the original cohort or the validation cohort. Randomization is based on the computer-generated random digits table. This study consists of two independent and consecutive stages:

1. Establishment and improvement of the HVPGBFM model: For 100 patients in the original cohort, biofluid mechanics specialists will use each patient's computed tomography, blood tests, Doppler ultrasound and HVPG results to adjust the parameters of the HVPGBFM model in order to make each patient's HVPGBFM and HVPG values match well.
2. Assessment of the HVPGBFM model: For 100 patients in the validation cohort, biofluid mechanics specialists will use each patient's computed tomography, blood tests and Doppler ultrasound results to calculate each patient's HVPGBFM according to the HVPGBFM model established previously. Biofluid mechanics specialists will make no changes to the HVPGBFM model and will have no access to patients' HVPG results in this cohort. Finally, the researchers will compare each patient's HVPGBFM and HVPG value and make an assessment of the HVPGBFM model.

Each patient's HVPG measurement will be performed after finishing computed tomography, blood tests and Doppler ultrasound. These results and other clinical data will be inaccessible to professionals for HVPG measurements in order to prevent certain biases. Each patient's computed tomography, blood tests, Doppler ultrasound and HVPG measurement will be performed within 30 days and treatments that may affect HVPG value will be avoided during this period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Patients with cirrhosis or portal hypertension, scheduled for HVPG measurement.

Exclusion Criteria:

* Female patients who are pregnant or nursing.
* Patients who are medically unstable, terminally or seriously ill, or patients whose clinical course is unpredictable.
* Patients with clinically unstable cardiac disease, for example: congenital heart defect, arrhythmia, uncontrolled heart failure (NYHA Class IV).
* Patients with respiratory distress syndrome or clinically unstable pulmonary disease, for example: pulmonary hypertension, pulmonary emboli, pulmonary vasculitis, emphysema.
* Patients with severe coagulation disorders.
* Patients with unstable occlusive disease or thrombosis within the hepatic, portal, or mesenteric veins.
* Patients who are allergic to iodinated contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between HVPGBFM and HVPG by Bland-Altman plot. | 7 days
  The numeric correlation between HVPGBFM and HVPG will be analysed by using Bland and Altman's limits of agreement analysis.
Correlation between HVPGBFM and HVPG by linear regression analysis. | 7 days
  The numeric relationship between HVPGBFM and HVPG will be analysed by using linear regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Luo, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin JY, Zhang CH, Zheng L, Li HJ, Zhu YM, Fan X, Li F, Xia Y, Huang MZ, Yang SH, Qi XL, Huo HZ, Chen HS, Lou XL, Luo M. Establishment and assessment of the hepatic venous pressure gradient using biofluid mechanics (HVPGBFM): protocol for a prospective, randomised, non-controlled, multicentre study. BMJ Open. 2019 Dec 3;9(12):e028518. doi: 10.1136/bmjopen-2018-028518. PMID 31796472

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03470389/Prot_SAP_001.pdf